CLINICAL TRIAL: NCT06147869
Title: Phonophoresis Versus Low-Level Laser Therapy on Dequervain Tenosynovitis After Delivery
Brief Title: Phonophoresis Versus Low-Level Laser on Dequervain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Reham Attia Mohamed Khotapy, student at master degree, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phonophoresis versus laser
Record Dates: First submitted 2023-11-09; First posted 2023-11-28 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: de Quervain Tenosynovitis
MeSH Terms: conditions — De Quervain Disease | interventions — Phonophoresis; Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: This study will be carried out on forty lactating women suffering from De Quervain's tenosynovitis after 6 weeks from the delivery. They will be selected randomly from the out patient clinic of orthopedic in Kasr El Aini Hospital. Their ages will be ranged from 25-35 years old, their body mass index (BMI) will not exceed 30 Kg/m2 and their parity will be ranged from (2-4 children).
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- photopheresis (Active Comparator)
  Interventions: Device: phonophoresis
- Low level laser (Active Comparator)
  Interventions: Device: Low level laser therapy

INTERVENTIONS:
Device: phonophoresis — Phonophoresis is a method of driving topically applied substances across tissues using ultrasound (US) to enhance percutaneous absorption of selected drugs such as corticosteroids, local anaesthetics, and salicylates
  Arms: photopheresis
Device: Low level laser therapy — Low-level laser (light) therapy (LLLT) is a fast-growing technology used to treat a multitude of conditions that require stimulation of healing, relief of pain and inflammation, and restoration of function.
  Arms: Low level laser

SUMMARY:
De Quervain's tenosynovitis is a frequently encountered pain of the hand and wrist. It results from compression and irritation of the extensor pollicis brevis and abductor pollicis longs tendons as they pass through the first dorsal compartment of the wrist. Patients complain of tenderness and swelling proximal to the radial styloid process, as well as pain in the wrist and on the radial side of the hand. Owing to persistent pain and inflammation, the pinch and grasp strength of the hand is considerably compromised, coupled with tenderness over the anatomical snuff box. Although the condition occurs in both females and males, it is significantly more common in women, especially during pregnancy and postpartum. This condition can be caused by micro traumas that occur in the course of repetitive mechanical activities and systemic diseases of the connective tissue.The symptom of de Quervain syndrome is pain in the forearm at the height of the radial styloid process. The pain intensifies during the extension of the thumb. Other symptoms include redness and swelling in the region. Physiotherapeutic treatment is an important element of conservative treatment of de Quervain syndrome .

DETAILED DESCRIPTION:
Phonophoresis is a method of driving topically applied substances across tissues using ultrasound (US) to enhance percutaneous absorption of selected drugs such as corticosteroids, local anaesthetics, and salicylates. Despite prevalent applications in various musculoskeletal conditions including de Quervain's disease, few modalities have been the target of as much controversy and speculation as phonophoresis. Standardised research is needed to accurately determine the efficacy of phonophoresis in pregnant females suffering from de Quervain's disease; more so because this vulnerable group is generally excluded from routine clinical trials and prevailing knowledge about the same is scant. Our study provides objective evidence regarding the applicability of phonophoresis in treating de Quervain's disease in pregnant women. It describes appropriate drug concentration, vehicle type, US frequency, and the mode for bringing about maximal improvements in the condition In physiotherapy LLLT is commonly used to relieve pain, reduce inflammation and accelerate tissue regeneration. So, it is usually recommended to treat De quervain's tenosynovitis, sprains, strains, low back pain, sciatica, postsurgical pain, shoulder pain, Sacro-iliac joint pain, Symphyseal pain, carpal tunnel syndrome, coccydynia, fibromyalgia, osteoarthritis, rheumatoid arthritis, disc herniation or degeneration, neuropathic pain, tendinitis, tennis elbow and plantar fasciitis. In the same time, according to The North American Association for Laser Therapy, LLLT is contraindicated in pregnancy, cancer, epileptic conditions and on eyes De Quervain's tenosynovitis is most common in women 30 to 50 years of age. Patients typically report several weeks of pain, often severe, on the radial aspect of the wrist at about the level of the radial styloid. Wrist pain and grip weakness are the hallmarks of de Quervain's tenosynovitis. Pinch grip, thumb extension or abduction. and wrist motion exacerbate and reproduce the pain.The pain of de Quervain's tenosynovitis can extend proximally up the forearm from the region of the anatomic "snuff box." Repetitive activities, especially activities that involve pinching with the thumb while moving the wrist in either the radial or ulnar direction, result in inflammation and pain within the shared tendon sheath of the abductor pollicis longus and extensor pollicis brevis

ELIGIBILITY:
Inclusion Criteria:

- 1. All participates are clinically diagnosed as they have De Quervain's tenosynovitis . 2. All patient will have positive Finkelstein test. 3. All patient will have severe pain, tenderness and swelling near the base of the thumb over the styloid process of the radius of their dominant hand and limitation of motion of the thumb and wrist joint. 4. Their ages will be ranged from 25-35 years old. 5. Their body mass index (BMI) will not exceed 30 kg/m2

* The type of delivery is normal and caesarean section.
* Their parity will be ranged from (2-4 children).
* All patients will not receive any medical treatment to relieve pain or decrease inflammation.
* All patients are not pregnant.

Exclusion Criteria:

* (1) Patients have diabetic mellitus, hypertension. (2) Patients have any cardiovascular diseases, heart diseases, renal diseases or any diseases (3) Patients have Rheumatoid Arthritis or Gout. (4) Patients have Cervical spondylosis with radiculopathy or any spinal diseases. (5) Patients have leukemia or tumor(benign or malignant)or even breast cancer. (6) Patients have double crush syndrome, carpal bone fracture or joint osteo-arthritis. (7) Patients have any deformities in their hands. (8) Patients have burns, ulcers, open wounds or any skin diseases in their dominant hands. (9) Patients have received medications or have injected with steroid in their tender point.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women with dequervain tenosynovities pospartum
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 4 weeks
  This scale will be used by each patient before and after the treatment course to estimate the intensity of pain. The Visual Analogue Scale (VAS) is a graphic rating scale with numerical values ranging from 0 to 4, placed equidistantly on a line 10 cm long, drawn horizontally.

CONTACTS AND LOCATIONS:
Locations (1):
- Sadat General Hospital, Cairo, Egypt